CLINICAL TRIAL: NCT04608019
Title: Streamlined Treatment of Pulmonary Exacerbations in Pediatrics (Pilot)
Brief Title: Streamlined Treatment of Pulmonary Exacerbations in Pediatrics Pilot Study
Acronym: STOP-PEDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington, the Collaborative Health Studies Coordinating Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP-PEDS
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; oral antibiotics; pulmonary exacerbation; pediatric
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Antibiotics (Experimental): increased airway clearance plus early initiation of oral antibiotics
  Interventions: Other: Immediate Antibiotics
- Tailored Therapy (Experimental): increased airway clearance alone, with addition of antibiotics for worsening symptoms or failure to improve
  Interventions: Other: Tailored Treatment

INTERVENTIONS:
Other: Immediate Antibiotics — increase airway clearance/start oral antibiotics right away
  Arms: Immediate Antibiotics
Other: Tailored Treatment — increase airway clearance and start oral antibiotics later if symptoms get worse or do not get better
  Arms: Tailored Therapy

SUMMARY:
STOP PEDS is a pilot study of children with CF ages 6-18 across 10 sites in North America. The primary goal is to assess the acceptability and feasibility of a multicenter randomized trial comparing immediate antibiotics versus tailored therapy for pulmonary exacerbation (PEx) treatment in this population.

DETAILED DESCRIPTION:
STOP PEDS is a pilot study of children with CF ages 6-18 across 10 sites in North America. The primary goal is to assess the acceptability and feasibility of a multicenter randomized trial comparing immediate antibiotics versus tailored therapy for pulmonary exacerbation (PEx) treatment in this population. The primary endpoint is the proportion of participants in the tailored arm who did not take any oral antibiotics in the 28 days following randomization.

Ultimately, we want to learn:

* What is the best way to treat pulmonary exacerbations?
* Should everyone with a pulmonary exacerbation take antibiotics?
* Do the benefits of starting antibiotics at the first signs of illness outweigh the possible risks, like side effects and antibiotic resistance?

This pilot study is designed to determine if an interventional study to help answer these questions is feasible. Up to 120 participants will be enrolled and followed through their well state of health, then for 28 days following their first randomized exacerbation. Enrollment will stop after 80 pulmonary exacerbation events have been randomized, even if this does not require 120 participants. Due to the nature of the study, the identity of treatment assignment will be known to investigators, research staff, and patients (ie, not blinded).

Total duration of this pilot study is expected to be approximately 18 months: 6 months for participant recruitment and 12 months for follow up. Participants could be monitored for up to 18 months if they do not have an exacerbation. However, it is anticipated that the majority of participants will experience a randomizable PEx event and therefore have a shorter follow up period.

ELIGIBILITY:
Enrollment Inclusion Criteria:

1. Age 6 to <19 years
2. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   1. sweat chloride ≥ 60 mEq/liter
   2. two disease-causing variants in the cystic fibrosis transmembrane conductive regulator (CFTR) gene
3. Written informed consent (and assent when applicable) obtained from participant or participant's legal representative and ability of participant to comply with the requirements of the study
4. Able to perform acceptable and reproducible spirometry
5. FEV1 ≥ 50% predicted at enrollment based on the Global lung Initiative (GLI) reference equations
6. At least 1 course of oral or IV antibiotics for respiratory symptoms since January 1, 2019.
7. Ability to receive text messages and access the internet

Enrollment Exclusion Criteria:

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
2. Previous randomization in the study
3. Receiving antibiotics for a PEx at the time of enrollment or within the 21 days prior to enrollment. Individuals may be re-screened ≥21 days after completion of antibiotics if they are at their baseline state of health, per self-report.
4. Treatment with systemic corticosteroids at enrollment. Individuals may be re- screened ≥21 days after completion of systemic corticosteroids if they are at their clinical baseline, per self-report.
5. History of solid organ transplant
6. History of positive culture for Mycobacterium abscessus in the 12 months prior to enrollment
7. Treatment with antibiotics for any non-tuberculous mycobacteria (NTM) at enrollment
8. Three or more IV antibiotic-treated PEx in the 12 months prior to enrollment
9. Treatment with chronic oral antibiotics other than azithromycin at enrollment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Delayed antibiotics | 28 days
  The proportion of participants in the tailored arm who did not take any oral antibiotics in the 28 days following randomization

SECONDARY OUTCOMES:
Consent | 6 months
  Proportion of approached patients consenting to enroll
Pulmonary Exacerbations Reported | 18 months
  Proportion of Pulmonary Exacerbations in which symptoms are reported within 7 days of onset
Randomization Criteria | 18 months
  Proportion of Pulmonary Exacerbation events meeting randomization criteria
Participant Exacerbations | 18 months
  Proportion of enrolled participants experiencing a randomizable Pulmonary Exacerbation
Randomized Exacerbations | 18 months
  Proportion of randomizable Pulmonary Exacerbations that undergo randomization
Day 28 Follow-up | 18 months
  Proportion of participants with a randomized Pulmonary Exacerbation that attends an in-person Day 28 follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Donald B. Sanders, MD, Principal Investigator — Riley Children's Hospital, Indianapolis, IN; Margaret Rosenfeld, MD, Principal Investigator — Seattle Children's Hospital, Seattle, WA
Locations (10):
- United States (10):
  - Tucson Cystic Fibrosis Center, Tucson, Arizona
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago & Northwestern University, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Texas Children's Hospital and Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley J, McAlister O, Elborn S. Pulmonary function, inflammation, exercise capacity and quality of life in cystic fibrosis. Eur Respir J. 2001 Apr;17(4):712-5. doi: 10.1183/09031936.01.17407120. PMID 11401068
- [Result] Sanders DB, Bartz TM, Zemanick ET, Hoppe JE, Hinckley Stukovsky KD, Cogen JD, Bendy L, McNamara S, Enright E, Kime NA, Kronmal RA, Edwards TC, Morgan WJ, Rosenfeld M. A Pilot Randomized Clinical Trial of Pediatric Cystic Fibrosis Pulmonary Exacerbations Treatment Strategies. Ann Am Thorac Soc. 2023 Dec;20(12):1769-1776. doi: 10.1513/AnnalsATS.202303-245OC. PMID 37683122
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37683122/